CLINICAL TRIAL: NCT04704804
Title: Feasibility of MRI Workflow Alone in External Radiotherapy for the Treatment of Brain and Prostate Tumors
Acronym: PRIS
Status: Completed | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-2020-09
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer; Brain Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prostate cancer: Man with cancer and localized (non-metastatic) prostate cancer
  Interventions: Diagnostic Test: Synthetic CT Scan
- Brain cancer: Male or Female with a brain tumor (primitive)
  Interventions: Diagnostic Test: Synthetic CT Scan

INTERVENTIONS:
Diagnostic Test: Synthetic CT Scan — method of generating CT-synthetic image from MRI

SUMMARY:
In radiotherapy, Magnetic Resonance Imaging (MRI) is used as a complement to the CT scanner because it provides better tissue contrast and therefore more precise delineations without the need for additional irradiation. However, MRI does not allow the definition of the electronic densities of the tissues necessary for dose calculation.

In this work, we sought to measure the feasibility of a method for generating CT-synthetic images from MRI in terms of dosimetric and geometrical precision for the purpose of MRI workflow alone (see diagram). The cerebral sphere and the prostate are the two tumor locations considered. All patients will have a planning CT (reference) and an MRI in the treatment position. The contours of the structures will be contoured by a radiotherapist on both the MRI and the reference CT. Synthetic CTs will be generated from the MRI with the method of automatic assignment of densities in five classes. The volumes bypassed and the dosimetries performed will be compared. A study of the quality of the images generated from MRI for dose calculation and images for the verification of per-treatment positioning will be performed.

DETAILED DESCRIPTION:
This is a prospective single-center dosimetry study that exhaustively included brain tumor and prostate cancer patients treated at the ICO Site d'Angers by external radiotherapy and prior to which they were given an MRI and a simulation CT in treatment position over a 12-month period.

For patients who agree to participate in the study, CT-synthetic images will be generated from the MRI images by automatic assignment of densities (5 classes).

Reference CT images from CT and synthetic CT images from MRI will be available for comparison for all eligible patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Male or Female with a (primary) brain tumour or Male with cancer and localized (non-metastatic) prostate cancer
3. Patient having benefited from a planning MRI scan in treatment position performed according to the new acquisition modalities (allowing the generation of CT-synthetics by automatic assignment of densities) performed since January 2020 and a planning scanner in treatment position prior to external radiotherapy.
4. Good general condition (SP < 3)

Exclusion Criteria:

1. Excluded forms of the disease,
2. MRI-specific contraindications (claustrophobia, foreign bodies)
3. Obesity preventing the placement of equipment (contention/antennae)
4. Poor general condition (SP > or = 2) preventing the patient from standing on the table -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with prostate or brain cancer receiving an MRI in addition to the simulated CT scan prior to the start of their external radiotherapy treatment
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
describe the differences in volumetric and dosimetric accuracy between potential planning from MRI alone by CT-synthetics generation and standard planning from CT | 3 month
  Comparison of the contours of target volumes and organs at risk and comparison of dose distributions (dosimetries)

SECONDARY OUTCOMES:
Measurement of the quality of images generated from MRI for dose calculation and images for verification of per-treatment positioning relative to the reference CT in an MRI-only workflow objective. | 3 month
  Comparison of CT-synthetic CT images generated from MRI to the reference CT and Comparison of shifts performed during patient repositioning

CONTACTS AND LOCATIONS:
Overall Officials: Damien AUTRET, Principal Investigator — INSTITUT DE CANCEROLOGIE DE L'OUEST
Locations (1):
- Institut de Cancerologie de L'Ouest, Angers, France

IPD SHARING:
Plan to Share IPD: No